CLINICAL TRIAL: NCT03885817
Title: Physically Active During Cancer Treatment
Brief Title: Physically Active During Cancer Treatment (FAKT)
Acronym: FAKT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Alesund Hospital (Other); Helse Nord-Trøndelag HF (Other); Ullevaal University Hospital (Other); Sorlandet Hospital HF (Other Government); Asker & Baerum Hospital (Other); Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015/1050
Record Dates: First submitted 2019-02-06; First posted 2019-03-22 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Neoplasms, Colorectal
Keywords: Exercise therapy; Fatigue; Adjuvant chemotherapy; Peripheral neuropathy, chemotherapy induced; Nutritional guide
MeSH Terms: conditions — Colorectal Neoplasms; Fatigue; Peripheral Nervous System Diseases | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise training and nutritional guide (Experimental): Standard recommendations regarding physical activity and nutrition. An individually tailored exercise program and nutritional guide during adjuvant chemotherapy.
  Interventions: Behavioral: Exercise training and nutritional guide; Other: Standard follow-up care
- Standard follow-up care (Active Comparator): Standard recommendations regarding physical activity and nutrition.
  Interventions: Other: Standard follow-up care

INTERVENTIONS:
Behavioral: Exercise training and nutritional guide — 30 minutes of a combination of sensorimotor- and strength training guided by a physical therapist twice a week. In addition 90 minutes a week of moderate intensity aerobic training or 45 minutes a week of high intensity aerobic training. Once a month the participants will fill out the form, PG-SGA SF, and he or she will be referred to a nutritionist if the score is 2 or higher. The intervention period lasts as long as the participants receives adjuvant chemotherapy, i.e. 3 - 6 months.
  Arms: Exercise training and nutritional guide
Other: Standard follow-up care — standard recommendations regarding physical activity and nutrition during the period with adjuvant chemotherapy.

SUMMARY:
This randomized controlled trial aims to investigate whether an individually tailored exercise program and nutritional guide can affect the development of self-reported peripheral sensory neuropathy and fatigue in patients with colorectal cancer receiving adjuvant chemotherapy.

DETAILED DESCRIPTION:
Colorectal cancer is the second most common cancer in Norway with 4332 new cases in 2017. Standard of care is radical surgery followed by adjuvant chemotherapy for some, depending on the stage of the disease. Most commonly, a combination of Oxaliplatin and Capecitabine or 5-fluorouracil is given for 3 to 6 months.

A common side effect of Oxaliplatin is peripheral sensory neuropathy, which occur in different degree in over 90 % of the patients. There is no established treatment to prevent or reduce Oxaliplatin induced peripheral neuropathy. A few minor studies have been published indicating that physical activity can reduce the patient's experience of chemotherapy-induced peripheral neuropathy.

Most patients receiving chemotherapy will experience fatigue in some degree. It has been shown in several studies that exercise can reduce cancer related fatigue, though most studies have been performed among women with breast cancer.

There are a limited number of randomized controlled clinical trials looking at the effects of physical exercise during ongoing adjuvant chemotherapy in colorectal cancer patients. Thus, there is a clear need for further studies on physical exercise in this patient group.

In the period from January 2017 to November 2018 the investigators did a non-randomized pilot study to test the feasibility of the exercise intervention in this patient group, and to calculate sample size for the randomized trial.

The 9-item European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) Chemotherapy Induced Peripheral Neuropathy (CIPN20) sensory subscale will be used to measure peripheral sensory neuropathy. Each item is rated on a scale from 1 ("not at all") to 4 ("very much"), and the total raw score ranges from 9 to 36. The raw scores will be linearly transformed to a 0 to 100 scale (higher scores represent worse CIPN severity). A difference of 10 is considered clinically significant. The sample size calculation is based on a two-sided t-test. Aim is to demonstrate a difference in patient-reported sensory peripheral neuropathy between the two groups 3 months after randomization. It is postulated that the intervention group develops less degree of peripheral sensory neuropathy than the control group. Based on the answers obtained from the questionnaire in the pilot study, a standard deviation (SD) of 12.5 is assumed for the change between baseline and 3 months. To detect a difference of 10 with a strength of 80% and with a significance level of 0.05, there should be 25 patients in each arm. A drop out of 20% is taken into account based on experience in the pilot study. This suggests that 64 patients should be included in this study.

Patients scheduled for adjuvant Oxaliplatin based combination chemotherapy will be recruited from cancer clinics in Norway, and randomized to an intervention group or a control group. Before randomization and start of the first cycle of chemotherapy, the study participants will perform baseline testing and fill in the different questionnaires.

The intervention with exercise training starts around the same time as adjuvant chemotherapy starts, usually 4 -6 weeks postoperatively, and lasts as long as the adjuvant treatment, i.e. 3 - 6 months. Participants start with an individual session with a physiotherapist at the hospital. A treadmill submaximal heart rate test is done to give the participants instructions regarding the recommended intensity zones during cardio training.

The exercise intervention consists of three components: sensorimotor training (SMT), strength exercises, and aerobic training. The SMT and strength exercises are carried out twice a week as guided training together with the physiotherapist, each session lasting 30 minutes. In addition, instruction is given to do minimum 90 minutes a week of moderate intensity (60 - 75 % of maximum heart rate) home-based aerobic training, or 45 minutes with high intensity (80 - 85 % of maximum heart rate) aerobic training.

Participants in the intervention group receive a pulse watch to guide the intensity of the aerobic exercise. The participants will register completed training in a training log. Based on previous experience with physical activity and exercise, individual guidance is provided.

Once a month participants will fill out the form, Patient-Generated Subjective Global Assessment Short Form (PG-SGA SF), and will be referred to a nutritionist if the score is 2 or higher. Regardless of the score on this form and group affiliation, participants may be referred to a nutritionist based on clinical judgment.

In the pilot study, also a qualitative study was carried out with semi-structured interviews evaluating patient's expectations and experiences regarding the physical exercise training. Depending on the information power obtained in the current sample, additional interviews of patients in this randomized trial might be done.

ELIGIBILITY:
Inclusion Criteria:

* Radical resection for colon- or rectal cancer past 3 months, and scheduled for adjuvant, Oxaliplatin-based, combination chemotherapy.
* Histologically confirmed adenocarcinoma.
* Able to read and understand Norwegian.
* Able to carry out the intervention.
* Performance Status (PS) 0 - 2.

Exclusion Criteria:

* Serious comorbidities that contraindicate physical exercise, based on the treating physician's assessment.
* Unable to give informed consent.
* Treated for other cancer last 5 years prior to inclusion (with the exceptions of basal cell carcinoma of the skin and carcinoma in situ in the cervix).
* Prior treatment with Oxaliplatin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Patient reported peripheral sensory neuropathy | Baseline to 3 months
  The 9-item European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) Chemotherapy Induced Peripheral Neuropathy (CIPN20) sensory subscale will be used to measure sensory neuropathy. Each item is rated on a scale from 1 ("not at all") to 4 ("very much"), and the total raw score ranges from 9 to 36. The raw scores will be linearly transformed to a 0 to 100 scale (higher scores represent worse CIPN severity).

SECONDARY OUTCOMES:
Fatigue | Baseline to 3, 6, 9, 12, 24 and 36 months
  Fatigue Questionnaire (FQ) will be used to measure fatigue. FQ contains 13 questions, is generic, and has well-documented psychometric properties. Each question is rated on a scale from 0 ("not at all" or "less than usual") to 3 ("much worse than usual"). FQ measures physical fatigue (PF) (seven questions, scores between 0-21) and mental fatigue (MF) (four questions, scores between 0-12). All questions are combined and constitute total fatigue (TF) (scores between 0-33) Higher scores indicate more fatigue.
Change in patient reported peripheral sensory neuropathy. | Baseline to 3, 6, 9, 12, 24 and 36 months
  European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) Chemotherapy Induced Peripheral Neuropathy (CIPN20) is a twenty questions quality-of-life questionnaire that has been developed to elicit patients' experience of symptoms and functional limitations related to CIPN (chemotherapy-induced peripheral neuropathy). CIPN20 has 3 sub-scales; a sensory, a motor and an autonomous. The sensory subscale has 9 items where each item is rated on a scale from 1 ("not at all") to 4 ("very much"), and the total raw score ranges from 9 to 36. The raw scores will be linearly transformed to a 0 to 100 scale (higher scores represent worse CIPN severity).
Change in patient reported motor neuropathy | Baseline to 3, 6, 9, 12, 24 and 36 months
  The 8-item European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) Chemotherapy Induced Peripheral Neuropathy (CIPN20) motor subscale will be used to measure motor neuropathy. Each item is rated on a scale from 1 ("not at all") to 4 ("very much"), and the total raw score ranges from 8 to 32. The raw scores will be linearly transformed to a 0 to 100 scale (higher scores represent worse CIPN severity).
Change in patient reported autonomic neuropathy | Baseline to 3, 6, 9, 12, 24 and 36 months
  The 3-item European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) Chemotherapy Induced Peripheral Neuropathy (CIPN20) autonomic subscale will be used to measure autonomic neuropathy. Each item is rated on a scale from 1 ("not at all") to 4 ("very much"), and the total raw score ranges from 3 to 12. The raw scores will be linearly transformed to a 0 to 100 scale (higher scores represent worse CIPN severity).
Clinicians reported neuropathy | Baseline to 3, 6 and 12 months.
  Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 will be used to grade neuropathy using the CTCAE terms Paresthesia (grade 1 -3), Peripheral sensory neuropathy (grade 1 - 4) and Peripheral motor neuropathy (grade 1 - 5). Grading will be performed at baseline, after 3 and 12 months for those who receives 3 months of adjuvant chemotherapy, and at baseline, after 3, 6 and 12 months for those who receives 6 months of adjuvant chemotherapy.
Change in body mass index (BMI) | Baseline to 3, 6 and 12 months.
  Weight and height will be combined to report BMI in kg/m^2. These measures will be taken at baseline, after 3 and 12 months for those who receives 3 months of adjuvant chemotherapy, and at baseline, after 3, 6 and 12 months for those who receives 6 months of adjuvant chemotherapy.
Change in systolic blood pressure (sBP) | Baseline to 3, 6 and 12 months.
  sBP is measured in mmHg (millimeter Mercury). This measure will be taken at baseline, after 3 and 12 months for those who receives 3 months of adjuvant chemotherapy, and at baseline, after 3, 6 and 12 months for those who receives 6 months of adjuvant chemotherapy.
Change in diastolic blood pressure (dBP) | Baseline to 3, 6 and 12 months.
  dBP is measured in mmHg (millimeter Mercury). This measure will be taken at baseline, after 3 and 12 months for those who receives 3 months of adjuvant chemotherapy, and at baseline, after 3, 6 and 12 months for those who receives 6 months of adjuvant chemotherapy.
Change in waist circumference. | Baseline to 3, 6 and 12 months.
  The waist circumference is measured when the patient is standing upright. Locate the midpoint between the lower rib and the top of the iliac crest and mark the point with a marker. Do not use the umbilicus as a measuring point. Place the tape measure on the mark. Ask the patient to hold the tape measure while walking around the patient. Check that the tape measure is horizontal in the middle of the back and that it lies against the body without tightening. Ask the patient to breathe out quietly. Read the circumference to the nearest 0.1 cm. Repeat the measurement and calculate the average.This measure will be taken at baseline, after 3 and 12 months for those who receives 3 months of adjuvant chemotherapy, and at baseline, after 3, 6 and 12 months for those who receives 6 months of adjuvant chemotherapy.
Change in HDL-cholesterol | Baseline to 3, 6 and 12 months.
  serum HDL-cholesterol (mmol/L). Blood analysis will be taken at baseline, after 3 and 12 months for those who receives 3 months of adjuvant chemotherapy, and at baseline, after 3, 6 and 12 months for those who receives 6 months of adjuvant chemotherapy.
Change in Triglycerides | Baseline to 3, 6 and 12 months.
  serum-triglycerides (mmol/L). Blood analysis will be taken at baseline, after 3 and 12 months for those who receives 3 months of adjuvant chemotherapy, and at baseline, after 3, 6 and 12 months for those who receives 6 months of adjuvant chemotherapy.
Change in Glycated hemoglobin (HbA1c) | Baseline to 3, 6 and 12 months.
  Blood HbA1c (mmol/mol). Blood analysis will be taken at baseline, after 3 and 12 months for those who receives 3 months of adjuvant chemotherapy, and at baseline, after 3, 6 and 12 months for those who receives 6 months of adjuvant chemotherapy.
Change in Glucose | Baseline to 3, 6 and 12 months.
  serum glucose (mmol/L). Fasting blood analysis will be taken at baseline, after 3 and 12 months for those who receives 3 months of adjuvant chemotherapy, and at baseline, after 3, 6 and 12 months for those who receives 6 months of adjuvant chemotherapy.
Change in Body Composition | Baseline to 3 and 12 months
  A Dexa Scan will be performed to evaluate change in Body Composition
Nutritional status | Baseline, 1, 2, 3, 4, 5 and 6 months
  At baseline and thereafter once a month until completion of adjuvant therapy, nutritional status is evaluated with the Patient-Generated Subjective Global Assessment Short Form (PG-SGA SF). This is a validated questionnaire, filled in by the patients to determine malnutrition status. The short form consists of four boxes with different questions. Box 1 is about weight and weight loss, and the score ranges from 0 - 5, where higher score indicates more weight loss. Box 2 is about food intake, and the score range is from 0 - 4, where higher score indicates more difficulties with food intake. Box 3 is about symptoms that have kept one from eating enough past two weeks. The score range is from 0 - 24, where higher score indicates more symptoms. Box 4 is about activities and function, and the score range is from 0 - 3, where higher score indicates a lower functional level.
Change in Quality Of Life: EORTC QLQ-C30 Version 3.0 | Baseline to 3, 6, 9, 12, 24 and 36 months
  The cancer-specific questionnaire European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTC QLQ-C30 Version 3.0) measures health-related quality of life. Participants rate the degree that each item has applied to them during the past week on a four-point Likert scale (1, not at all; 4, very much). The average of the item scores gives a raw score, and the raw score will be transformed to a 0 to 100 scale. Higher scores indicate higher QOL.
Completion of adjuvant treatment 1 | 3 to 6 months
  At the end of adjuvant treatment, the percentage given by Oxaliplatin relative to the calculated full dose is calculated (%)
Completion of adjuvant treatment 2 | 3 to 6 months
  At the end of adjuvant treatment, the percentage given by Fluorouracil or Capecitabine relative to the calculated full dose is calculated (%)
Completion of adjuvant treatment 3 | 3 to 6 months
  At the end of adjuvant treatment,the total number of days the treatment courses have been delayed are calculated (days).
Physical capacity | Baseline to 3, 6 and 12 months.
  The submaximal exercise test, "Modified Shuttle Walk Test", is used to measure physical capacity. The test is performed three times in those who receives 3 months of adjuvant chemotherapy (baseline, 3 and 12 months), and four times in those who receives 6 months of adjuvant chemotherapy (baseline, 3, 6 and 12 months).
Self-reported physical activity | Baseline to 3, 6, 9, 12, 24 and 36 months
  Self-reported physical activity is measured using three questions from the Health Survey in Nord-Trøndelag (HUNT) which include frequency, duration and intensity of physical activity.
Muscle strength | Baseline to 3, 6 and 12 months.
  Strength of the lower limbs is indirectly measured by the test "Sit to Stand" which records how many times the patient is able to stand up and sit down from a chair within 30 seconds. This is measured three times for those who receives 3 months of adjuvant chemotherapy (baseline, 3 and 12 months). This is measured four times for those who receives 6 months of adjuvant chemotherapy (baseline, 3, 6 and 12 months).
Balance 1 | Baseline to 3, 6 and 12 months.
  Balance is measured with the test "Tandem standing". The test is performed with both closed and open eyes, and measures how many seconds (up to a maximum of 30 seconds), one can stand in the tandem position. The test is performed three times in those who receives 3 months of adjuvant chemotherapy (baseline, 3 and 12 months), and four times in those who receives 6 months of adjuvant chemotherapy (baseline, 3, 6 and 12 months).
Balance 2 | Baseline to 3, 6 and 12 months.
  Balance is measured with the test "Standing balance on one and one leg". The test is performed with both closed and open eyes, and measures how many seconds (up to a maximum of 30 seconds), one can stand on one leg. The test is performed three times in those who receives 3 months of adjuvant chemotherapy (baseline, 3 and 12 months), and four times in those who receives 6 months of adjuvant chemotherapy (baseline, 3, 6 and 12 months).
Haematological toxicity | Baseline to 6 months.
  Using Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0, all grade 3 or more events for platelet- or neutrophil count will be registered. In addition, all admissions to hospital due to febrile neutropenia will be registered.
Time before return to work | Baseline to 3, 6, 9, 12, 24 and 36 months
  The rate of sick leave is recorded at baseline and every 3 months up to one year after inclusion using a questionnaire. This is also recorded after 2 and 3 years, using the same questionnaire.
Overall- and disease free survival | Baseline to 5 years
  Time of recurrence or death is recorded by annual journal review for up to 5 years after inclusion. This is defined as time from randomization to respectively recurrence or death.

OTHER OUTCOMES:
Serious adverse events (SAE) | Baseline to 6 months
  All serious events that may be related to the intervention will be recorded.
Patient's expectations and experiences | Baseline, 3 and 6 months
  Semi-structured interviews
Medical treatment for hypertension. | Baseline, 3, 6 and 12 months
  It will be registered whether the patient receives medical treatment for hypertension, and is answered with "yes" or "no". This will be recorded at baseline, after 3 and 12 months for those who receives 3 months of adjuvant chemotherapy, and at baseline, after 3, 6 and 12 months for those who receives 6 months of adjuvant chemotherapy.
Diagnosed with type 2 diabetes. | Baseline, 3, 6 and 12 months
  It will be registered whether the patient is diagnosed With type 2 diabetes , and is answered with "yes" or "no". This will be recorded at baseline, after 3 and 12 months for those who receives 3 months of adjuvant chemotherapy, and at baseline, after 3, 6 and 12 months for those who receives 6 months of adjuvant chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Arne Solberg, md phd, Study Director — St. Olavs Hospital
Locations (5):
- Norway (5):
  - Ålesund sjukehus, Ålesund
  - Sørlandet sykehus, Kristiansand, Kristiansand
  - Levanger sykehus, Levanger
  - Ullevål, Oslo
  - Kreftklinikken, St Olavs Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hatlevoll I, Oldervoll LM, Wibe A, Stene GB, Stafne SN, Hofsli E. Physical exercise during adjuvant chemotherapy for colorectal cancer-a non-randomized feasibility study. Support Care Cancer. 2021 Jun;29(6):2993-3008. doi: 10.1007/s00520-020-05789-z. Epub 2020 Oct 8. PMID 33030598